CLINICAL TRIAL: NCT04179149
Title: Enriched Environments: a Multi-level Integrative Medicine Intervention for Endometriosis
Brief Title: Enriched Environments in Endometriosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ponce Medical School Foundation, Inc. (Industry)
Collaborators: University of Oxford (Other); DHR Health Institute for Research and Development (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1R21HD098481-01 (NIH)
Record Dates: First submitted 2019-10-07; First posted 2019-11-27 (Actual); Results first posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Endometriosis-related Pain; Endometriosis; Pelvic Pain; Quality of Life; Inflammation Pelvic
Keywords: endometriosis; chronic pelvic pain; quality of life; inflammation; stress
MeSH Terms: conditions — Endometriosis; Pelvic Pain; Pelvic Inflammatory Disease; Inflammation

STUDY DESIGN:
Intervention Model Description: In this RCT study, subjects randomized to the intervention condition will receive the Environmental Enrichment (EE) intervention as an adjuvant to standard gynecological care consisting of hormonal, analgesic or surgical treatment as necessary according to their symptoms during the study period. Participants randomized to the control condition will receive only standard care as necessary according to their symptoms during the study period in addition to an online patient training online seminar.
Who Masked: Outcomes Assessor
Masking Description: Investigators will not be blinded because the two arms are receiving different interventions. However, data will be coded such that data entry and initial analysis can be done in a blinded fashion as to intervention group until ad hoc analysis are conducted.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Environmental enrichment (Experimental): Subjects randomized to the intervention condition will receive the environmental enrichment intervention (social support, open spaces, novel stress relief activities) as an adjuvant to standard gynecological care consisting of hormonal, analgesic or surgical treatment as necessary according to their symptoms during the study period.
  Interventions: Behavioral: Environmental enrichment
- Controls (No Intervention): Participants randomized to the control condition will receive only standard care as necessary according to their symptoms during the study period plus an online patient training module.

INTERVENTIONS:
Behavioral: Environmental enrichment — The experimental group will participate in six modules that mimic and integrate the three hallmarks of environmental enrichment: social interaction (more animals per cage = support group meetings, online support), novelty (toys and activities = exposure to new hands-on activities), and larger enclosures (larger cages = meetings in open environments). There will be 2 interventions per month, for three months, and a follow up 3 months after the end of the intervention
  Arms: Environmental enrichment

SUMMARY:
The investigators propose to conduct a randomized behavioral trial that will produce a clinically useful multi-level integrative medicine model to be used in stress- and inflammation-related disorders that can easily be implemented with current pharmacological interventions to alleviate pain and improve QoL.

DETAILED DESCRIPTION:
Endometriosis is a chronic inflammatory and painful condition that affects 176 million women in their reproductive years worldwide, and has substantial costs related to health care and loss in work productivity. The symptoms of endometriosis-chronic, incapacitating pain and infertility-cause high levels of stress, leading to poor quality of life (QoL) in affected women. Stress is known to affect the physiology of pelvic organs and to disturb the hypothalamic-pituitary-adrenal (HPA) axis leading to chronic, painful, inflammatory disorders. The team has documented a relationship between stress, HPA dysregulation and endometriosis. In an animal model the team demonstrated that stress exacerbates disease manifestations whereas the ability to control the level of stress results in smaller lesions and less inflammation. Further, the team has identified social support as one of the parameters that most significantly impacts QoL in women with endometriosis. Environmental enrichment (EE) can produce beneficial effects in models of chronic diseases improving anxiety and immune-related disturbances, and can block the effects of chronic stress on brain hippocampal integrity. The team recently found that EE can effectively minimize lesion size and numbers, and also decreased anxiety in this animal model. Together, these data support the basic premise of this proposal: EE interventions can overcome chronic stress thus reversing the negative influences on mental health status (depression/anxiety levels), inflammation/HPA axis (inflammatory cytokines, cortisol), and clinical course (pain levels) of endometriosis, leading to improved QoL. The central objective of this study is to refine and test a multi-modal intervention based on the EE paradigm tested in our animal model and translated it to the human scenario, to produce data on its effectiveness. The team hypothesizes that the EE interventions can be effectively adapted for women with endometriosis resulting in pain reduction and improved QoL. To test our hypothesis, our multidisciplinary team with combined expertise in endometriosis, psychology, physiology, neuroscience, gynecology, and stress management has adapted the experimental EE model to the human scenario. By applying a combined approach (systematic review of the literature, and input from a patient advisory committee) the team has developed six EE modules to be tested in human subjects. This study consists of two specific aims. In aim 1, the team will assess feasibility and acceptability of the EE interventions through a collaborative approach involving a patient population to refine EE modules. Under aim 2, the team will conduct a randomized clinical trial (RCT) of the EE intervention to determine its efficacy in improvement of pelvic pain and QoL (primary outcomes), and inflammation, HPA axis disturbances, and mental health (depression, anxiety) (secondary outcomes), measured before and after the intervention. With this purpose, the team will use a case control study design for the RCT where cases will receive the intervention as an adjuvant to standard gynecologic care for endometriosis, while controls will receive standard of care only. The proposed work will produce a clinically useful multi-level integrative medicine model to be used in stress- and inflammation-related disorders that can easily be implemented with current pharmacological interventions to alleviate pain and improve QoL.

ELIGIBILITY:
Inclusion Criteria:

* premenopausal adult women
* adults 18 and 49 y/o
* diagnosed with endometriosis by surgery
* symptomatic
* refractory to hormonal treatment
* able to provide written informed consent

Exclusion Criteria:

* Pregnant women (or who become pregnant during the study period)
* Asymptomatic
* Documented visual, cognitive or physical impairment that would interfere with participation or consent.
* Currently under mental health pharmacological treatment
* Currently using steroid medications.
* Diagnosis of pain syndromes (e.g., fibromyalgia, chronic fatigue syndrome).

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2019-09-13 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Idhaliz Flores, PhD, Principal Investigator — Ponce Medical School Foundation
Locations (1):
- Ponce Medical School Foundation, Ponce, PR, Puerto Rico

IPD SHARING:
Plan to Share IPD: No
At this point, no individual patient data will be made available to other investigators

REFERENCES:
- [Result] Nieves-Vazquez CI, Detres-Marquez AC, Torres-Reveron A, Appleyard CB, Llorens-De Jesus AP, Resto IN, Lopez-Rodriguez V, Ramos-Echevarria PM, Castro EM, Flores I. Feasibility and acceptability of an adapted environmental enrichment intervention for endometriosis: A pilot study. Front Glob Womens Health. 2023 Jan 4;3:1058559. doi: 10.3389/fgwh.2022.1058559. eCollection 2022. PMID 36683601
- [Result] De Hoyos G, Ramos-Sostre D, Torres-Reveron A, Barros-Cartagena B, Lopez-Rodriguez V, Nieves-Vazquez C, Santiago-Saavedra F, Appleyard CB, Castro EM, Flores I. Efficacy of an environmental enrichment intervention for endometriosis: a pilot study. Front Psychol. 2023 Oct 10;14:1225790. doi: 10.3389/fpsyg.2023.1225790. eCollection 2023. PMID 37885745

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We completed recruitment for both study cohorts of cases and controls. We started patient recruitment in September 2019 via a social media campaign and regular media (newspaper articles, radio, TV). Printed flyers and posters were distributed among local gynecology offices. Our targeted recruitment was 60 subjects per study group or 120 subjects total for both sessions. By the start of the study we recruited 29 patients in the intervention group and 27 in the control group.
Groups:
- Environmental Enrichment: Subjects randomized to the intervention condition will receive the Environmental Enrichment (EE) intervention (social support, open spaces, novel stress relief activities) as an adjuvant to standard gynecological care consisting of hormonal, analgesic or surgical treatment as necessary according to their symptoms during the study period.
  Environmental enrichment: The experimental group will participate in six modules that mimic and integrate the three hallmarks of Environmental Enrichment: social interaction (more animals per cage = support group meetings, online support), novelty (toys and activities = exposure to new hands-on activities), and larger enclosures (larger cages = meetings in open environments). There will be 2 interventions per month, for three months, and a follow up 3 months after the end of the intervention
- Controls: Participants randomized to the control condition will receive only standard care as necessary according to their symptoms during the study period in addition on participation in an online patient training module.
Period: Overall Study
Arm/Group | Environmental Enrichment | Controls
Started | 29 | 27
Completed | 12 | 27
Not Completed | 17 | 0

BASELINE CHARACTERISTICS:
Groups:
- Environmental Enrichment: Subjects randomized to the intervention condition will receive the EE intervention (social support, open spaces, novel stress relief activities) as an adjuvant to standard gynecological care consisting of hormonal, analgesic or surgical treatment as necessary according to their symptoms during the study period.
  Environmental enrichment: The experimental group will participate in six modules that mimic and integrate the three hallmarks of EE: social interaction (more animals per cage = support group meetings, online support), novelty (toys and activities = exposure to new hands-on activities), and larger enclosures (larger cages = meetings in open environments). There will be 2 interventions per month, for three months, and a follow up 3 months after the end of the intervention
- Controls: Participants randomized to the control condition will receive only standard care as necessary according to their symptoms during the study period PLUS an online patient training module. They were visited by members of the study team twice at their homes or preset meeting place to obtain samples and surveys.
- Total: Total of all reporting groups
Arm/Group | Environmental Enrichment | Controls | Total
Number analyzed (Participants) | 29 | 27 | 56
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 29 | 27 | 56
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.7 (6.677) | 34.0 (7.638) | 33.34 (7.123)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 27 | 56
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 29 | 27 | 56
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 29 | 27 | 56
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Puerto Rico | 29 | 27 | 56
pelvic pain [Count of Participants; unit: Participants] | 29 | 25 | 54
Dyspareunia [Count of Participants; unit: Participants] | 22 | 20 | 42
Baseline pelvic pain levels [Mean (Standard Deviation); unit: units on a scale] — The Numerical Pain Scale (NRS) is a self-reported scale of pain ranging from 1 to 10, 1 being no pain, and 10 being the worst imaginable pain. Scale: 1-4 mild pain, 5-7 moderate pain, 8-10 severe pain
  units on a scale | 8 (2.2) | 6.4 (3.3) | 7.2 (2.9)
Perceived stress (PSS14) [Mean (Standard Deviation); unit: units on a scale] — Perceived Stress Scale 14 or PSS14:
  PSS-14 scores are obtained by reversing the scores on the seven positive items, e.g., 0=4, 1=3, 2=2, etc., and then summing across all 14 items. Items 4, 5, 6, 7, 9, 10, and 13 are the positively stated items. Individual scores on the PSS can range from 0 to 40 with higher scores indicating higher perceived • stress. ► Scores ranging from 0-13 would be considered low stress. ► Scores ranging from 14-26 would be considered moderate stress. ► Scores ranging from 27-40 would be considered high perceived stress.
  units on a scale | 32.5 (5.7) | 28.0 (4.4) | 30.3 (5.6)

OUTCOME MEASURES:

1. Primary Outcome: Pain Perception
Description: Mean level of maximum pain using the Visual Analog Scale (VAS), in which 1 is no pain and 10 is the worst pain imaginable. Categories: 1-4 low pain; 5-7 moderate pain; 8-10 severe pain. Therefore, the higher the score in the VAS the higher the pain level.
Time Frame: at baseline, at end of the intervention and 3 months after the end of intervention
Population: The total of participants is not equal to the total number of participants enrolled because not all participants completed this particular questionnaire of the several instruments they had to complete.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Environmental Enrichment | Controls
Number analyzed (Participants) | 27 | 22
units on a scale
  Baseline | 7.0 (2.8) | 6.2 (3.4)
  End of intervention | 7.2 (1.7) | 5.1 (3.0)
  3-months after | 6.3 (2.4) | 6.6 (2.5)

2. Primary Outcome: Quality of Life (QoL)
Description: QoL global impact scores measured using the Endometriosis Health Profile 30 (EHP-30), a disease-specific questionnaire to measure health related quality of life. The EHP-30 was developed by Jones et al., in 2001. Part 1 The first part contains 30 questions relevant to all women with endometriosis covering five areas: pain, emotional well-being, control and powerlessness, social support and self imaging scales. Each domain score is calculated by dividing the total scores of each item in the domain by the maximum possible score of all items in the domain multiplied by 100. Our outcome of interest is the global impact score, calculated as the mean of all completed subscale scores, with a range of 0 to 100. The global impact score ranges from 0 (indicating the best health status) to 100 (indicating the worst health status). No subscales are reported.
Time Frame: at baseline, at end of the intervention and 3 months after the end of intervention (for intervention); at baseline and end of intervention (for controls)
Population: The total of participants is not equal to the total number of participants enrolled because not all participants completed this particular questionnaire out of the many instruments that they needed to complete; also not all completed the Follow up End of intervention questionnaire in the control group (16 out of 19 participants).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Environmental Enrichment | Controls
Number analyzed (Participants) | 26 | 19
score on a scale
  Baseline | 61.0 (13.5) | 60.1 (18)
  End of intervention: number analyzed (Participants) | 26 | 16
  End of intervention | 56.6 (16.0) | 56.2 (11.5)
  3-months after: number analyzed (Participants) | 11 | 0
  3-months after | 50.9 (11.0) |

3. Secondary Outcome: Perceived Stress Levels 14
Description: Perceived stress levels will be measured using the Perceived Stress Scale 14 at baseline, end of interventions and 3 months from the end of intervention for the intervention group, but only at baseline and end of the intervention for the control group. The survey asks the following 14 questions about stressful situations and helps determine what stress is to the participant and how stressful they feel their life to be. Higher scores indicate higher levels of stress.
  The 14 items are scored from 0 to 4. Total scores range from 0 to 56. Score categories are:
  Low Stress (scores 0 - 18) Moderate Stress (scores 19 - 37) High Stress (scores 38 - 56)
Time Frame: at baseline, at end of the intervention and 3 months after the end of intervention (for the intervention); at baseline and end of the intervention (for controls)
Population: The total of participants is not equal to the total number of participants enrolled because not all participants completed this particular questionnaire out of the many instruments they were asked to complete.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Environmental Enrichment | Controls
Number analyzed (Participants) | 27 | 22
score on a scale
  Baseline | 30.0 (5.8) | 28.8 (5.8)
  End of intervention | 28.2 (5.3) | 27.5 (6.1)
  3 months after: number analyzed (Participants) | 17 | 0
  3 months after | 25.7 (5.3) |

4. Secondary Outcome: Depressive Symptomatology
Description: The Patient Health Questionnaire-8 (PHQ-8) is a validated self-report tool used to assess the severity of depressive symptoms over the previous two weeks. The PHQ-8 includes 8 items, each scored on a 4-point scale:
  0 = Not at all
  1. = Several days
  2. = More than half the days
  3. = Nearly every day Total score range: 0 to 24 Directionality: Higher scores indicate greater depressive symptom severity (i.e., worse outcomes).
  Interpretation of total scores:
  0-4: None to minimal depression 5-9: Mild depression 10-14: Moderate depression 15-19: Moderately severe depression 20-24: Severe depression The PHQ-8 was assessed at baseline, immediately post-intervention, and at 3-month follow-up for the intervention group, and at baseline and post-intervention for the control group.
Time Frame: at baseline, at end of the intervention and 3 months after the end of intervention; and at baseline and post-intervention for the control group.
Population: The total of participants is not equal to the total number of participants enrolled because not all participants completed this particular questionnaire out of the many instruments they were asked to complete; also not all participants completed the follow up questionnaires at the end of the intervention or at 3 months after (only for the intervention group)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Environmental Enrichment | Controls
Number analyzed (Participants) | 29 | 27
score on a scale
  Baseline | 10.8 (4.5) | 11.3 (5.9)
  End of intervention | 9.0 (4.7) | 8.9 (5.2)
  3 months after: number analyzed (Participants) | 20 | 0
  3 months after | 6.9 (4.0) |

5. Secondary Outcome: Anxiety Symptomatology
Description: General Anxiety Disorder 7 (GAD-7) survey assessed at baseline, end of intervention and 3 months from the end of intervention. The GAD-7 scores were also represented with clinical categorizations of anxiety levels as follows: GAD-7 score of 0-4 (none), 5-9 (mild), 10-14 (moderate), and 15-21 (severe).
Time Frame: at baseline, at end of the intervention and 3 months after the end of intervention (for the intervention group) and at baseline and end of the intervention (for the control group)
Population: The total of participants is not equal to the total number of participants enrolled because not all participants completed this particular questionnaire out of many instruments they were asked to complete.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Environmental Enrichment | Controls
Number analyzed (Participants) | 29 | 27
score on a scale
  Baseline | 11.7 (4.7) | 10.9 (6.2)
  End of intervention | 8.9 (4.2) | 10.1 (6.6)
  3 months after: number analyzed (Participants) | 20 | 0
  3 months after | 6.9 (4.1) |

ADVERSE EVENTS:
Time Frame: Six (6) months
Description: Definition of adverse events is in accord with the clinical trials website guidelines.
Arm/Group | Environmental Enrichment | Controls
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/27
Other Adverse Events (participants affected / at risk) | 1/29 | 0/27
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Environmental Enrichment (N=29) | Controls (N=27)
skin reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — A mild and transient irritation to an essential oil was reported by one participant during the aromatherapy session.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-11-15): https://cdn.clinicaltrials.gov/large-docs/49/NCT04179149/Prot_SAP_000.pdf
  • Informed Consent Form (2019-07-08): https://cdn.clinicaltrials.gov/large-docs/49/NCT04179149/ICF_001.pdf